CLINICAL TRIAL: NCT05885074
Title: Mechanistic Insights to Weight Loss Maintenance Through SGLT2 Inhibitors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 300011125
Record Dates: First submitted 2023-05-11; First posted 2023-06-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin Arm (Experimental): Investigator will enroll 12 obese participants who have intentionally lost greater than or equal to 5% of body weight through a non-pharmacological structured weight loss program based on diet and exercise within the last 6 months. The participants will take empagliflozin 25mg/day orally for 12 months.
  Interventions: Drug: Empagliflozin Arm; Other: Exercise capacity VO2 maximum determination; Other: Exercise Challenge
- Placebo Arm (Placebo Comparator): Investigator will enroll 12 obese participants who have intentionally lost greater than or equal to 5% of body weight through a non-pharmacological structured weight loss program based on diet and exercise within the last 6 months. The participants will take a placebo pill orally once a day for 12 months.
  Interventions: Other: Control Arm; Other: Exercise capacity VO2 maximum determination; Other: Exercise Challenge

INTERVENTIONS:
Drug: Empagliflozin Arm — The subject will be randomized, in a double-blind manner to Empagliflozin 25mg once daily for a period of 12 months
  Arms: Empagliflozin Arm
Other: Control Arm — The subject will be randomized, in a double-blind manner to receive placebo once daily for a period of 12 months
  Arms: Placebo Arm
Other: Exercise capacity VO2 maximum determination — Each participant's maximal oxygen capacity will be determined using a modified Bruce treadmill protocol and will also undergo a DEXA scan to determine the body mass.
Other: Exercise Challenge — Each participant will walk at 70 % of his/her VO2max for 20 minutes on treadmill and will also undergo a resting energy expenditure test.

SUMMARY:
Obesity increases the risk of cardiometabolic diseases such as hypertension and diabetes. Weight loss interventions such as low-calorie diet and physical activity are effective for weight loss in the short term, but weight loss maintenance (WLM) with low-calorie diet and physical activity is challenging. Weight loss is associated with a reduction in the amount of calories needed to maintain the body at rest, called the resting energy expenditure (REE), which may be a probable mechanism for this lack of WLM. Most individuals are unable to adequately change their diet and increase their physical activity levels to overcome this decrease in REE which prevents WLM. Therefore, techniques that increase REE may promote WLM in these individuals. Pre-clinical studies for Empagliflozin - Sodium-glucose Cotransporter-2 (SGLT2) inhibitor have shown an increase in REE. Thus, in addition to reducing the cardiovascular risk, SGLT2 inhibitor may promote WLM by increasing REE. This study aims to promote WLM in obese individuals by increasing the REE using SGLT2 inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 years
* Body mass index more than or equal to 30 kg/m2 who have lost ≥5% of body weight within the past 6 months without taking any pharmacotherapy for weight loss

Exclusion Criteria:

* Age less than 18 years at screening.
* Untreated systolic BP <100 or >160 mmHg at baseline, or diastolic BP <80 or >100 mmHg at baseline
* Women who are pregnant or breastfeeding or who can become pregnant and not practicing an acceptable method of birth control during the study (including abstinence)
* Taking pharmacotherapy indicated for weight loss, such as GLP-1 agonists or with weight loss as an adverse event
* History of Type I Diabetes
* History of lung disease
* Have any past or present illness of cardiovascular disease, including myocardial infarction, angina, cardiac arrhythmia, diabetes, stroke, TIA, or seizure
* Current or past (<12 months) history of smoking
* Estimated glomerular filtration rate (GFR) < 60 ml/min/1.73 m2 (CKD-EPI equation) urine albumin creatinine ratio ≥30 mg/g
* Hepatic Transaminase (AST and ALT) levels >3x the upper limit of normal
* Significant psychiatric illness
* Anemia (men, Hct < 38%; women, Hct <36%)
* Inability to exercise on a treadmill
* Consumption of more than 2 alcoholic drinks daily
* Any contraindications to empagliflozin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Resting Energy Expenditure | 12 months
  Change in Resting Energy Expenditure between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention

SECONDARY OUTCOMES:
Change in Body Weight | 12 months
  Change in Body Weight between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in Body Mass Index | 12 months
  Change in Body Mass Index between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in Waist Circumference | 12 months
  Change in Waist Circumference between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in HbA1C levels | 12 months
  Change in HbA1C levels between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in lipid profile | 12 months
  Change in Lipid profile between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in HOMA-IR | 12 months
  Change in HOMA-IR between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in ESR | 12 months
  Change in ESR between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in CRP | 12 months
  Change in CRP between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in IL-6 | 12 months
  Change in IL-6 between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in TNF-α | 12 months
  Change in TNF-α between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in glucagon-like peptide-1 (GLP-1) | 12 months
  Change in glucagon-like peptide-1 (GLP-1) between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in peptide YY (PYY) | 12 months
  Change in peptide YY (PYY) between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in ghrelin | 12 months
  Change in ghrelin between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in glucose-dependent insulinotropic polypeptide (GIP) | 12 months
  Change in glucose-dependent insulinotropic polypeptide (GIP) between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention
Change in glucagon | 12 months
  Change in glucagon between the two arms (Empagliflozin v/s Placebo) from baseline and after 12 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided